CLINICAL TRIAL: NCT04090047
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE 2-PERIOD STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSES OF ITRACONAZOLE ON THE PHARMACOKINETICS OF A SINGLE DOSE OF PF-06700841 IN HEALTHY PARTICIPANTS
Brief Title: A Study to Investigate the Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of PF-06700841 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7931033
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Heathy Participants
MeSH Terms: interventions — PF-06700841; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06700841 and Itraconazole (Experimental): This fixed sequence, 2-period arm will consist of two treatments. Participants will receive a single oral dose of 30 milligrams (mg) PF-06700841 on Day 1 in Period 1. On Days 1-7 in Period 2, Itraconazole 200mg will be administered once daily(QD). On Day 4 of Period 2, co-administration of Itraconazole 200 mg and 30 mg PF-06700841 tablets will occur.
  Interventions: Drug: PF-06700841; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-06700841 — PF-06700841 oral tablets in 5mg and 25mg provided for a 30mg dose
Drug: Itraconazole — 200 mg oral solution administered as 20 milliliters(mL) (10 mg/mL)
  Other Names: Sporanox®

SUMMARY:
An open-label, fixed-sequence, 2-period study to investigate the effect of multiple oral doses of itraconazole on a single oral dose of PF-06700841 PK in healthy participants. The study will consist of two treatment periods in one fixed sequence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, full physical examination, which includes blood pressure (BP) and pulse rate measurement, clinical laboratory tests, and 12-lead ECG.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
* Participant with a history of known hypersensitivity to itraconazole or its excipients or to other azole antifungals.
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B core antibody (HBcAb), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON®- tuberculosis (TB) Gold or equivalent test.
* Have a history of any lymphoproliferative disorder (such as Epstein Barr Virus [EBV] related lymphoproliferative disorder, as reported in some participants on other immunosuppressive drugs), history of lymphoma, leukemia, myeloproliferative disorders, multiple myeloma, or signs and symptoms suggestive of current lymphatic disease.
* Have or have had clinically significant infections within the past 3 months prior to the first dose of investigational product (eg, those requiring hospitalization or parenteral antibiotics, or as judged by the Investigator), evidence of any infection within the past 7 days prior to the first dose of investigational product, herpes simplex within 12 weeks or history of disseminated herpes simplex infection, symptomatic herpes zoster or recurrent (>1 episode) or disseminated herpes zoster.
* Have undergone significant trauma or major surgery within 4 weeks of Screening.
* Have been vaccinated with live or attenuated live vaccine within the 6 weeks prior to the first dose of investigational product, or expects to be vaccinated with these vaccines during study treatment, or within the 6 weeks following the last dose of investigational product.Recombinant subunit vaccines (eg, Shingrix®) are permitted and it is preferable that the last dose is administered at least 4 weeks prior to Day 1.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Female participants taking hormone replacement therapy within 28 days prior to the first dose of study treatment.
* A positive urine drug test.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Use of tobacco/nicotine containing products in excess of 5 cigarettes/day.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Female participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 60 days after the last dose of itraconazole.
* Female nursing participants will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measured concentration (AUClast) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUCinf) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Maximum Observed Plasma Concentration (Cmax) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) | screening to last phone all follow up
  For male and women of non-childbearing potential (WONCBP), last phone call follow up is 28-35 days after last dose For women of childbearing potential (WOCBP), last phone call follow up is 60-65 days after last dose
Incidence of Serious Adverse Events(SAE), and AEs leading to Discontinuation | screening to last phone call follow up
  For male and women of non-childbearing potential (WONCBP), last phone call follow up is 28-35 days after last dose For women of childbearing potential (WOCBP), last phone call follow up is 60-65 days after last dose
The incidence of clinically significant abnormalities in vital signs | screening, pre-dose and 3 hours post-dose on Day 1 in Period 1; Pre-dose on Day 1, 3 hours post-dose on Day 4 and prior to discharge on Day 7 in Period 2
The incidence of clinically significant abnormalities in electrocardiograms(ECG) | screening, pre-dose and 3 hours post-dose on Day 1 in Period 1; Pre-dose on Day 1, 3 hours post-dose on Day 4 and prior to discharge on Day 7 in Period 2
The incidence of clinically significant abnormalities in clinical laboratory values | screening, Day -1 in Period 1 and prior to discharge in Period 2
Maximum plasma concentration(Cmax) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Plasma (Tmax) time to reach Cmax of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Terminal elimination half-life (t1/2) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Apparent clearance (CL/F) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Apparent volume of distribution(Vz/F) of PF-06700841 | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Maximum plasma concentration(Cmax) of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Plasma (Tmax) time to reach Cmax of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Area under the plasma concentration-time curve from time zero to the last measured concentration (AUClast) of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Metabolite/parent ratio (M/P) of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
Area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUCinf) of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
  if data permit
Terminal elimination half-life (t1/2) of PF-06700841 major metabolite (M1) | Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 in periods 1 and 2. Hour 72 in period 2
  if data permit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931033